CLINICAL TRIAL: NCT03251326
Title: Effects of Nabilone on Trauma Related Cue Reactivity in Cannabis Users With PTSD
Brief Title: Nabilone in Cannabis Users With PTSD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Margaret Haney, Professor of Neurobiology (in Psychiatry) at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 6971; U54DA037842 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: Cannabis; Post Traumatic Stress Disorder
MeSH Terms: conditions — Marijuana Abuse; Stress Disorders, Post-Traumatic | interventions — nabilone; nabiximols; Propranolol

STUDY DESIGN:
Intervention Model Description: All patients will contribute to each of 4 drug conditions (placebo, nabilone, smoked cannabis, and propranolol).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nabilone (Experimental): Nabilone capsules (4 mg)
  Interventions: Drug: Nabilone
- Propranolol (Active Comparator): Propranolol capsules (40mg)
  Interventions: Drug: Propranolol
- Smoked cannabis (Experimental): (0.0 and 5.6% THC)
  Interventions: Drug: Cannabis
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — Nabilone capsules (4 mg)
  Arms: Nabilone
Drug: Cannabis — Cigarettes (0.0 and 5.6% THC)
  Arms: Smoked cannabis
Drug: Propranolol — Propranolol capsules (40mg)
  Arms: Propranolol
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
Despite the prevalence of cannabis use among the PTSD population and self-reports that it is used to help cope with PTSD symptoms, the direct effects of cannabis on PTSD symptomology are unknown. The purpose of this placebo-controlled, within-subject study is to assess the effects of smoked cannabis and orally administered nabilone, a synthetic analog of THC, the primary psychoactive component of cannabis on multiple dimensions of PTSD symptomatology in cannabis smokers with PTSD.

DETAILED DESCRIPTION:
This study will compare the effects of smoked cannabis and nabilone on attentional bias toward trauma- related stimuli, subjective and emotional processing to a range of trauma-and non-trauma-related images and physiological reactivity to these stimuli in individuals with CUD and PTSD. Importantly, this study will also probe the abuse related potential of nabilone compared to smoked cannabis in this population, a critical aspect in determining the potential feasibility for its use clinically to treat CUD in PTSD populations. The effects of nabilone will be compared to propranolol as a positive control.

ELIGIBILITY:
Inclusion Criteria:

* Current cannabis use
* PTSD symptoms
* Able to give informed consent and comply with study procedures
* Women who are normally cycling and practicing an effective form of birth control other than hormonal contraceptives

Exclusion Criteria:

* Meeting criteria for certain current psychiatric disorders
* Clinical laboratory tests outside of normal limits
* History of clinically significant cardiac or respiratory diagnoses
* Current parole or probation
* Women who are currently pregnant or breastfeeding

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated and the PI and the study team left the institution; as such, no outcome data is available.
Groups:
- Active Nab > Plac Prop > Plac Cann: Nabilone capsules (4 mg) Propranolol placebo capsules (0 mg) Placebo cannabis (0.0% THC)
- Plac Nab > Act Prop > Plac Cann: Nabilone placebo capsules (0 mg) Propranolol capsules (40mg) Placebo cannabis (0.0% THC)
- Plac Nab > Plac Prop > Act Cann: Nabilone placebo capsules (0 mg) Propranolol placebo capsules (0 mg) Smoked cannabis (5.6% THC)
- Plac Nab > Plac Prop > Plac Cann: Nabilone placebo capsules (0 mg) Propranolol placebo capsules (0 mg) Placebo cannabis (0.0% THC)
Period: Overall Study
Arm/Group | Active Nab > Plac Prop > Plac Cann | Plac Nab > Act Prop > Plac Cann | Plac Nab > Plac Prop > Act Cann | Plac Nab > Plac Prop > Plac Cann
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Nabilone/Propranolol/Placebo + Smoked Cannabis/Placebo Placebo: Nabilone capsules (4 mg) Propranolol (40mg) Placebo (0mg nabilone or propranolol) Placebo cannabis (0.0% THC) Smoked cannabis (5.6% THC)
Arm/Group | Nabilone/Propranolol/Placebo + Smoked Cannabis/Placebo Placebo
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Cue Reactivity (Emotional Stroop Task)
Description: We cannot provide data as the study was terminated due to lack of feasibility. The staff responsible for data collection, organization, and cleaning have left the institution; we have made every effort to locate the data for the two participants who completed the study, but have been unsuccessful. We do not have access to the data.
Time Frame: 1 month
Population: We cannot provide data as the study was terminated due to lack of feasibility. The staff responsible for data collection, organization, and cleaning have left the institution; we have made every effort to locate the data for the two participants who completed the study, but have been unsuccessful. We do not have access to the data.
Arm/Group | Active Nab > Plac Prop > Plac Cann | Plac Nab > Act Prop > Plac Cann | Plac Nab > Plac Prop > Act Cann | Plac Nab > Plac Prop > Plac Cann
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (October 2015 - June 2019). Each participant's was enrolled in the study for approximately 1.5 months, during which adverse event data was collected (baseline through each of 4 experimental sessions).
Description: We cannot provide data as the study was terminated due to lack of feasibility. The staff responsible for data collection, organization, and cleaning have left the institution; we have made every effort to locate the data for the two participants who completed the study, but have been unsuccessful. We do not have access to the data.
Arm/Group | Active Nab > Plac Prop > Plac Cann | Plac Nab > Act Prop > Plac Cann | Plac Nab > Plac Prop > Act Cann | Plac Nab > Plac Prop > Plac Cann
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT03251326/Prot_000.pdf